CLINICAL TRIAL: NCT00688766
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study Evaluating the Efficacy and Safety of IPI-504 in Patients With Metastatic and/or Unresectable GIST Following Failure of at Least Imatinib and Sunitinib
Brief Title: Study Evaluating IPI-504 in Patients With Gastrointestinal Stromal Tumors (GIST) Following Failure of at Least Imatinib and Sunitinib
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on Independent Data Monitoring Committee (IDMC) recommendation.
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Collaborators: MedImmune LLC (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPI-504-06
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: GIST; Metastatic and/or Unresectable Gastrointestinal Stromal
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — tanespimycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IPI-504 (Experimental): retaspimycin hydrochloride (IPI-504) plus best supportive care
  Interventions: Drug: retaspimycin hydrochloride (IPI-504); Other: Best supportive care
- Placebo (Placebo Comparator): Placebo plus best supportive care
  Interventions: Drug: placebo; Other: Best supportive care

INTERVENTIONS:
Drug: retaspimycin hydrochloride (IPI-504) — IPI-504 is a novel small molecule inhibitor of heat shock protein 90 (Hsp90). Patients will receive 400 mg/m2 of IPI-504 as a 30-minute IV infusion twice weekly for 2 weeks followed by 1 week off.
  Arms: IPI-504
Drug: placebo — Patients will receive a 30-minute IV infusion twice weekly for 2 weeks followed by 1 week off.
  Arms: Placebo
Other: Best supportive care — Best supportive care will be according to institutional standard, but will not include administration of systemic cancer-specific therapies including chemotherapies, biologic therapies, investigational therapies, TKIs (e.g., imatinib, sunitinib, nilotinib, dasatinib), or local therapies such as surgery, radiotherapy, or lesion ablative therapies.

SUMMARY:
IPI-504-06 is a Phase 3, randomized, double-blind, placebo-controlled, multi-center study to evaluate the efficacy and safety of IPI-504 as compared to placebo in patients with metastatic and/or unresectable GIST following failure of at least imatinib and sunitinib.

Approximately 195 patients will be randomized using a 2:1 ratio to receive either IPI-504 (N=130) or placebo (N=65). Upon unblinding, patients receiving either IPI-504 or placebo may receive IPI-504 in the open-label portion of the study if defined inclusion criteria are met.

Early and frequent imaging timepoints (Weeks 2, 5, 8, 14 and every 6 weeks thereafter) are incorporated into this study to capture progression events and limit patient exposure to ineffective agents.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of study randomization.
* Histologically confirmed metastatic and/or unresectable GIST.
* Measurable disease on CT or MRI as defined by RECIST.
* Documented radiographic progression or intolerance to imatinib and sunitinib.
* Clinical failure of the most recent prior therapy for GIST. Note: There is no limit to the number of prior therapies a patient may have received.
* Eastern Cooperative Oncology Group (ECOG) performance status: 0 or 1.
* Hemoglobin ≥ 8.0 g/dL (80 g/L).
* Absolute Neutrophil Count ≥ 1500/µL (1.5 x 109/L).
* Platelets ≥ 100,000 /µL (100 x 109/L).
* ALT and AST ≤ 2.5 x upper limit of normal (ULN), or ≤ 5.0 x ULN if considered secondary to liver metastases.
* Alkaline phosphatase ≤ 2.5 x ULN, or ≤ 5.0 x ULN if considered secondary to liver metastases.
* Serum bilirubin ≤ 1.5 x ULN.
* PT and PTT ≤ 1.5 x ULN unless the patient is receiving warfarin. If the patient is receiving warfarin, the INR must be within therapeutic range.
* Serum creatinine ≤ 1.5 x ULN.

Exclusion Criteria:

* Previous administration of other known heat shock protein 90 (Hsp90) inhibitors.
* Surgery, radiotherapy, or lesion ablative procedure to the only area of measurable disease.
* Initiation or discontinuation of concurrent medication that is a potent CYP3A inhibitor less than 2 weeks prior to administration of IPI-504 or placebo.
* History of any of the following within the last 6 months: cardiac disease such as acute coronary syndrome or unstable angina, symptomatic congestive heart failure, uncontrolled hypertension, cirrhotic liver disease, cerebrovascular accident, or any other significant co-morbid condition or disease which, in the judgment of the investigator, would place the patient at undue risk or interfere with the study.
* Grade 3 or 4 hemorrhagic event within the last 6 months.
* Known human immunodeficiency virus positivity.
* Sinus bradycardia (resting heart rate < 50 bpm) secondary to intrinsic conduction system disease.
* QTcF ≥ 470 milliseconds, or previous history of clinically significant QTc prolongation while taking other medications.
* History of prior malignancies within the past 3 years other than non-melanomatous skin cancers that have been controlled, prostate cancer that has been treated and has not recurred, non-muscle-invasive bladder cancer, and carcinoma in situ of the cervix.
* Active or recent history (within 3 months) of keratitis or keratoconjunctivitis confirmed by ophthalmology or optometry exam.
* Presence of Left Bundle Branch Block, Right Bundle Branch Block plus left anterior hemiblock, bifascicular block, or 3rd degree heart block. This does not include patients with a history of these events with adequate control by pacemaker.
* Known CNS metastases.
* Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Compare the progression free survival (PFS) in both study arms | Multiple timepoints

SECONDARY OUTCOMES:
Compare the disease control rate (DCR) in both arms | Multiple timepoints
Compare the time to progression (TTP) in both arms | Multiple timepoints
Compare the overall survival (OS) in both arms | Continuous
Evaluate the safety and tolerability of IPI-504 in this patient population | Signing of the informed consent to 30 days after discontinuation of drug

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Santabarbara, M.D., Study Director — Infinity Pharmaceuticals, Inc.; George Demetri, MD, Principal Investigator — Dana-Farber Cancer Institute

REFERENCES:
- See also: Gist Support International - Patient Advocacy Group — http://www.gistsupport.org
- See also: The Liferaft Group - Patient Advocacy Group — http://www.liferaftgroup.org